CLINICAL TRIAL: NCT02042846
Title: Prospective Clinical Evaluation of the Bioabsorbable SportWelding FijiAnchor® for Ligament Repair of the Hand and Hand Wrist
Brief Title: Clinical Evaluation of the SportWelding FijiAnchor® in Hand and Hand Wrist Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SportWelding GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Spo-01
Record Dates: First submitted 2014-01-09; First posted 2014-01-23 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Lesion of Ligament of Wrist and/or Hand

ARMS (1):
- SportWelding Fiji Anchor (Experimental)
  Interventions: Device: SportWelding Fiji Anchor

INTERVENTIONS:
Device: SportWelding Fiji Anchor

SUMMARY:
The SportWelding FijiAnchor is an absorbable suture anchor which is inserted by applying ultrasonic energy. This provides an intimate bond between implant and bone delivering immediate stability.

The purpose of this study is to evaluate the surgical and clinical outcome of the SportWelding Fiji Anchor in ligament repair of the hand and hand wrist.

ELIGIBILITY:
Inclusion Criteria:

* Having a condition requiring (re)fixation or (re)construction of ligaments in the hand or hand wrist
* Being able to comprehend, sign, and date the written informed consent form (ICF)); and
* Being able to visit the hospital to be examined the repaired region after the procedure.

Exclusion Criteria:

* Having serious concomitant disease
* Being pregnant
* Having the control hand not suitable to serve as comparator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Operation success | Day 1
  Technical success confirmed at the end of surgery by mean of an assessment form (e.g anchor insertion without breaking and suture without pulling off from the tissue during surgery).
Procedure success | 12 weeks
  No dislodged/broken anchor nor ruptured sutures observed at 2, 6 and 12 weeks post operative evaluation

SECONDARY OUTCOMES:
Clinical function | 3 and 6 months
  Dash (Disabilities of the Arm, Shoulder and Hand) Score, PRWE (Patient-Related-Wrist-Evaluation) Score and strength of the operated and the non-operated control hand will be recorded after 6 and 12 months.
Adverse events | From Day 1 to 12 months
  All adverse events will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Arora, MD, Principal Investigator — Univ.-Klinik für Unfallchirurgie Innsbruck, Austria
Locations (1):
- Univ.-Klinik für Unfallchirurgie, Innsbruck, Tyrol, Austria